CLINICAL TRIAL: NCT06834178
Title: Hepatitis Elimination And Liver Care in South-East Austria (HEAL-S)
Brief Title: Non-interventional Study to Assess the Number of People With Untreated/Unknown HBV + HDV and HCV in South-East Austria
Acronym: HEAL-S
Status: Not yet recruiting | Type: Observational
Sponsor: Vanessa Stadlbauer-Koellner, MD (Other)
Collaborators: Medical University of Graz (Other)
Responsible Party: Sponsor-Investigator, Vanessa Stadlbauer-Koellner, MD, Univ. Prof. Dr. Vanessa Stadlbauer-Köllner, Medical University of Graz
Organization: Medical University of Graz (Other)
Other Study IDs: 1173/2024
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: HBV; HCV; HDV; Coinfection; Hepatitis B Coinfection; Hepatitis B
Keywords: HBV; HCV; HDV; Hepatitis B and D coinfection; untreated hepatitis; Hepatitis B; Hepatitis C; Hepatitis treatment
MeSH Terms: conditions — Coinfection; Hepatitis B; Hepatitis C

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HCV Cohort: Patients in the HCV cohort will be invited to laboratory evaluation. Patient visits correspond to routine and are not specific to the study - they include platelet count, liver biochemistry tests, virologic parameters (HCV, HIV, HBV), liver stiffness measurement using elastography (Fibroscan®, Echosens, France), counselling regarding HCV transmission and persons in whom plasma HCV RNA is detectable will be offered treatment with direct-acting antivirals (DAAs). The choice of DAA will be made according to individual comorbidities, comedications, previous HCV treatments, prescriber and personal preferences. Routine surveillance data under DAA treatment will be recorded. SVR is defined as HCV RNA not detectable after the end of DAA treatment. Furthermore, the suspected route of HCV transmission will be documented.
- HBV Cohort: In the HBV cohort, patients with missing or positive but untreated HDV serology and with positive HBV viral load and negative HDV serology, but no evidence of linkage to care will be contacted via telephone or mail and invited for evaluation as described above and linked to care including treatment of HBV infection according to the applicable clinical practice guidelines as well as prescriber and personal preferences.
  In case of positive HDV serology, HDV RNA testing will be performed and depending on the result, treatment of HBV/HDV coinfection will be initiated according to the applicable clinical practice guidelines as well as prescriber and personal preferences. Furthermore, the suspected route of HBV/HDV transmission will be assessed. Patient visit is part of routine treatment and done according to the respective treatment guidelines and the requirements of health insurance policy.

SUMMARY:
The HEAL-S study is a non-interventional study with retrospective data analysis. It consists of two parts. First a retrospective analysis based on nucleic acid testing (NAT) results will be performed. Two cohorts (HCV) and (HBV) will be established. Patients falling into one (or both) of the two cohorts will be invited to a prospective linkage-to-care study. In this part, patients are invited to the clinic, where the possibility of hepatitis treatment will be discussed.

DETAILED DESCRIPTION:
We hypothesize that in South-East Austria, a relevant number of persons are unaware of their HCV infection or their HDV status in case of HBV coinfection and therefore not yet sufficiently linked to care.

The study consists of two parts:

1. First a retrospective analysis based on nucleic acid testing (NAT) results will be performed: all results for HCV-RNA and HBV-DNA + HDV serology results obtained from the specific laboratories of the Diagnostic and Research Institute of Hygiene, Microbiology and Environmental Medicine between January 01, 2014 to December 31, 2023 will be retrieved through the laboratory information system. In the extracted dataset we will first verify that patients are alive and have a valid SVNR in Austria. Eligible patients (estimated 800) will be manually checked in our electronic patient record system (openMEDOCS) to verify that the patients had not been treated for HCV infection any time or lack HDV testing in case of HBV coinfection. The remaining patients comprise the target population.
2. Two cohorts (HCV) and (HBV) will be established. Patients falling into one (or both) of the two cohorts will be invited to a prospective linkage-to-care study. The patients from the target population will be contacted via telephone or mail and invited for assessment at Medical University of Graz. Numbers and percentages of persons called, reached, clinically assessed, treated, and cured (sustained virological response, SVR) will be evaluated.

2.1. HCV cohort Patients in the HCV cohort will be invited to laboratory evaluation. Patient visits correspond to routine and are not specific to the study - they include platelet count, liver biochemistry tests, virologic parameters (HCV, HIV, HBV), liver stiffness measurement using elastography (Fibroscan®, Echosens, France), counselling regarding HCV transmission and persons in whom plasma HCV RNA is detectable will be offered treatment with direct-acting antivirals (DAAs). The choice of DAA will be made according to individual comorbidities, comedications, previous HCV treatments, prescriber and personal preferences. Routine surveillance data under DAA treatment will be recorded. SVR is defined as HCV RNA not detectable after the end of DAA treatment. Furthermore, the suspected route of HCV transmission will be documented.

2.2. HBV cohort In the HBV cohort, patients with missing or positive but untreated HDV serology and with positive HBV viral load and negative HDV serology, but no evidence of linkage to care will be contacted via telephone or mail and invited for evaluation as described above and linked to care including treatment of HBV infection according to the applicable clinical practice guidelines as well as prescriber and personal preferences.

In case of positive HDV serology, HDV RNA testing will be performed and depending on the result, treatment of HBV/HDV coinfection will be initiated according to the applicable clinical practice guidelines as well as prescriber and personal preferences. Furthermore, the suspected route of HBV/HDV transmission will be assessed. Patient visit is part of routine treatment and done according to the respective treatment guidelines and the requirements of health insurance policy.

The active study participation ends with the linkage-to-care. The treatment of the viral hepatitis infection is not part of the study any more. The outcome of therapy will be assessed via chart review in retrospect.

ELIGIBILITY:
Inclusion Criteria:

* The target population for the HCV cohort consists of individuals with detectable plasma HCV RNA at the latest observation.
* The target population for the HBV cohort consists of individuals with detectable plasma HBV RNA at any time and no recorded HDV testing or a positive HDV serology.

Exclusion Criteria:

* No valid SVRN (german: Sozialversicherungsnummer, english: Social insurance number)
* No contact details available
* Documented Sustained Virological Response (HCV cohort)
* Documented assessment of HDV status (HBV cohort)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female patients in South-East Austria with undiagnosed HCV infection or with unknown HDV status in case of HBV infection.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of HCV patients that can be linked to care | 10/2024 - 10/2026
  To identify patients with detectable plasma HCV-RNA and subsequently treat them (HCV cohort)
Number of HDV patients that can be linked to care | 10/2024 - 10/2026
  To identify patients with HDV infection and link them to care (HBV/HDV cohort)

SECONDARY OUTCOMES:
Virological response (SVR) rate | 10/2024 - 10/2026
  To assess the sustained virological response (SVR) rate in this macroelimination program
Prevalence of HCV, HBV and HDV infection in South-East Austria | 10/2024 - 10/2026
  To estimate the prevalence of HCV, HBV and HDV infection in South-East Austria
Number of South-East Austria HCV patients treated since DAA treatment has been available | 10/2024 - 10/2026
  To estimate the number of South-East Austrian HCV patients treated since DAA treatment has been available
Number of HCV re-infections | 10/2024 - 10/2026
  To estimate the number of HCV re-infections
Number of patients with HBV infection who were not tested for HDV infection | 10/2024 - 10/2026
  To estimate the diagnostic gap in patients with HBV infection who were not tested for HDV infection
Number of patients with HBV infection who were not tested for HDV infection | 10/2024 - 10/2026
Number of HBV patients with HDV infection | 10/2024 - 10/2026

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Stadlbauer-Köllner, Univ. Prof. Dr., Principal Investigator — Medical University of Graz, Department of Gastroenterology and Hepatology, Medical University of Graz; Harald H. Kessler, Univ. Prof. Dr., Study Director — Diagnostic and Research Institute of Hygiene, Microbiology and Environmental Medicine, Medical University of Graz
Locations (1):
- Department of Internal Medicine, Division of Gastroenterology and Hepatology, Graz, Styra, Austria

IPD SHARING:
Plan to Share IPD: Undecided